CLINICAL TRIAL: NCT04018456
Title: Regenerative Root Canal Treatment of Mature Teeth With Pulp Necrosis and Apical Periodontitis Using Biodentine Compared With MTA: Randomized Clinical Double-blind Trial
Brief Title: Regenerative Endodontic Treatment of Mature Necrotic Teeth With Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amatallah Hussein Nasser Al-Rawhani, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CU-2019-7-7
Record Dates: First submitted 2019-07-07; First posted 2019-07-12 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Necrotic Pulp; Apical Periodontitis
Keywords: Necrotic pulp,; Apical periodontitis; Regeneration; MTA; Biodentine
MeSH Terms: conditions — Dental Pulp Necrosis; Periapical Periodontitis | interventions — tricalcium silicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants/ outcome assessor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodentine (Experimental): Intervention group: application of biodentine as pulp space barrier during regenerative endodontic treatment.
  Interventions: Other: Biodentine
- White MTA (Active Comparator): Control group: application of White MTA as pulp space barrier during regenerative endodontic treatment.
  Interventions: Other: White MTA

INTERVENTIONS:
Other: Biodentine — Biodentine is calcium silicate based cement which is bioactive and inductive material. Biodentine will be applied as coronal plug material.
  Arms: Biodentine
Other: White MTA — MTA is calcium silicate based cement which is bioactive and inductive material. MTA is used in most cases of regenerative endodontics and it will be applied as coronal plug material.
  Other Names: white mineral trioxide aggregate
  Arms: White MTA

SUMMARY:
The aim of this prospective, randomized, controlled double-blind study is to evaluate the effectiveness of biodentine compared with MTA used as pulp space barrier on discoloration of teeth after regenerative based non-obturation root canal treatment in mature single canal with pulp necrosis and apical periodontitis.

DETAILED DESCRIPTION:
• Regenerative endodontic treatment will be performed through two visits: First visit aims to clean and disinfect the tooth canal by copious irrigation with NaOCL and EDTA solution . At the end of first visit, canal will be dressed by CaOH as intracanal medicaments.

Second visit will be after two weeks. After removal of CaOH dressing by copius irrigation, evoking bleeding inside canal by over instrumentation. When blood become semi-coagulated, according to the random sequence number of the participants, either biodentine or white MTA will be placed as pulp space barrier.

At the end of treatment, the access cavity will be sealed with composite restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Tooth type: single-rooted teeth (anterior or premolar) encasing of one root canal with mature root (closed apex).
2. Negative response of pulp tissue to electrical or thermal pulp tester.
3. Widening in lamina dura or periapical radiolucency not more than 3 mm.

Exclusion Criteria:

* 1. Patients having significant systemic disorder or immunocompromised patients. 2. Teeth with generalized chronic periodontitis or have periodontal pocket larger than 3 mm.

  3. Teeth with developmental anomalies (i.e, dens invaginatusor a palatogingival groove).

  4. Teeth with previous root canal. 5. Teeth need to post and core as final restoration

Ages: 10 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Discoloration of teeth | Up to one Year after completion of regenerative endodontic treatment
  Discoloration of teeth that will be assessed clinically through follow up period 3, 6, 9, 12 months by visual examination and by using color shade guide (Tetric N shade guide, Ivoclar Vivadent) whether tooth discolored or not in comparison with the original preoperative color shade.

SECONDARY OUTCOMES:
Healing of Periapical Tissue | after 3, 6,9 and Up to 12 months after completion of regenerative endodontic treatment
  Healing of periapical tissue will be assessed clinically and radiographically through follow up period: 3, 6, 9, 12 months. When the case is clinically asymptomatic: (without sinus tract, swelling, with no palpation, or percussions pain) and radiographically showed absence or reduction of the radiolucency are together will considered successful of regenerative treatment.
Restoring the sensibility of tooth | after 6,9 and Up to 12 months after completion of regenerative endodontic treatment
  Electric pulp tester (EPT)

CONTACTS AND LOCATIONS:
Overall Officials: Amatallah HN Al-Rawhani, Master, Principal Investigator — Cairo University
Locations (1):
- Dentistry Faculty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arslan H, Ahmed HMA, Sahin Y, Doganay Yildiz E, Gundogdu EC, Guven Y, Khalilov R. Regenerative Endodontic Procedures in Necrotic Mature Teeth with Periapical Radiolucencies: A Preliminary Randomized Clinical Study. J Endod. 2019 Jul;45(7):863-872. doi: 10.1016/j.joen.2019.04.005. Epub 2019 May 31. PMID 31155298